CLINICAL TRIAL: NCT02808689
Title: Functional Medicine in Asthma (FAst) Study
Acronym: FAst
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FAst
Record Dates: First submitted 2016-06-16; First posted 2016-06-22 (Estimated); Last update posted 2021-04-01 (Actual); Status verified 2020-11

CONDITIONS: Asthma
Keywords: Moderate; Severe
MeSH Terms: conditions — Asthma; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Asthma Center (Active Comparator): Use of Currently Accepted Asthma Care Guidelines:
  1. Assessment and monitoring: the use of objective measures of lung function to assess severity of asthma and to monitor the course of therapy,
  2. Control of factors contributing to symptom exacerbation: environmental control measures to avoid or eliminate factors that precipitate asthma symptoms or exacerbations,
  3. Pharmacotherapy: comprehensive pharmacologic therapy for long-term management, and
  4. Education for partnership in care: patient education that fosters a partnership among the patient, his/her family, and clinicians.
  Interventions: Other: Currently Accepted Asthma Care Guidelines
- Asthma Center plus Functional Medicine (Active Comparator): All the factors in the Asthma Center Arm plus:
  Address lifestyle factors such as nutrition and exercise that influence long-term health and chronic diseases. The intention is to reduce ongoing biologic imbalances from deficiencies in dietary oxidants/antioxidants via vitamin supplementation, hormonal imbalances through evaluation and management, and the need for medications with unwarranted side effects that compound the chronic medical conditions and adverse effects (e.g. excess use of antibiotics), and to systematically evaluate intolerances to certain foods and additives.
  Interventions: Behavioral: Lifestyle Factors; Other: Customized use of Dietary Supplements

INTERVENTIONS:
Behavioral: Lifestyle Factors — Will look at nutrition and exercise that influence long-term health and chronic diseases.
  Arms: Asthma Center plus Functional Medicine
Other: Customized use of Dietary Supplements — Reduce ongoing biologic imbalances from deficiencies in dietary oxidants/ antioxidants via vitamin supplementation. Approach is customized based on results for laboratory testing.
  Arms: Asthma Center plus Functional Medicine
Other: Currently Accepted Asthma Care Guidelines — Use of asthma care guidelines set forth by the National Institutes of Health/National Heart, Lung and Blood Institute (NIH/NHLBI) and Global Initiative for Asthma
  Arms: Asthma Center

SUMMARY:
This is a pilot, proof of concept, early stage study. The study goal is to determine whether the Functional Medicine approach to the treatment of moderate to severe persistent asthma enhances standard guideline-based care with respect to asthma outcomes.

DETAILED DESCRIPTION:
Functional Medicine is a holistic approach to treating chronic conditions by attempting to address the underlying causes of chronic disease states. The purpose is to address the whole person, not just a set of symptoms. The patient care involves evaluating the interactions among genetic, in-utero, and lifetime environmental exposures. In addition, Functional Medicine specialists also aggressively address lifestyle factors such as nutrition and exercise that influence long-term health and chronic diseases. By doing so, the intention is to reduce ongoing biologic imbalances from deficiencies in dietary oxidants/antioxidants via vitamin supplementation, hormonal imbalances through evaluation and management, and the need for medications with unwarranted side effects that compound the chronic medical conditions and adverse effects (e.g. excess use of antibiotics), and to systematically evaluate intolerances to certain foods and additives.

Collaborating with Functional Medicine directly addresses the Guideline focus on control of factors contributing to symptom exacerbation as well as the Cleveland Clinic care path initiative goals of improving patient satisfaction with collaborative healthcare teams to modify risk factors and counsel on environmental/lifestyle modifications. This study will look at the effectiveness of adding a Functional Medicine approach to patient asthma care.

The investigators intention with this pilot study is to study subjective areas of medicine (symptoms and quality of life) as objectively as possible, in order to supplement asthma care guidelines with potential evidence of asthma-related quality of life, lung function/asthma control, and biomarker-based reduction of inflammation and improvement of immune status. Certainly there is value to both approaches and the aspects that are valuable need to be determined so that these two disciplines can have a more integrated approach moving forward and benefit a larger population in innovative and scientifically proven ways.

ELIGIBILITY:
Inclusion Criteria:

* Women and men with ages >18 and <65
* Nonsmokers or Former smokers quit >1 yr ago, with 15 pack-years or less history of smoking
* Clinical history consistent with moderate to severe asthma
* Measures of airflow obstruction and reactivity consistent with asthma (12% BD response and/or positive methacholine challenge test) historically or at initial/screening visit FEV1 between 40-100% predicted post bronchodilator
* Uncontrolled Asthma categorized ACT ≤19 (i.e. Not well controlled ACT= 16-19, Very Poorly Controlled ACT ≤ 15)
* Willing to be seen in Asthma Center and willing to consider Functional Medicine approach as an add-on to Asthma Center care
* Able to attend study visits as outlined in protocol.

Exclusion Criteria:

* Current smoker
* Life threatening asthma defined as 2 or more intubations for asthma in last 12 months
* Major psychiatric disturbance
* Any disorder, including but not limited to gastrointestinal, renal, neurological, infectious, endocrine, metabolic or other physical impairment, that is not stable in the opinion of the investigator
* Clinically important pulmonary disease other than asthma, including but not limited to COPD, pulmonary fibrosis, cystic fibrosis, bronchiectasis
* Pregnant or breastfeeding
* Controlled asthma defined by stability and by ACT >19 and physician discretion for 2-3 months
* Current asthma exacerbations, (exacerbations are defined by urgent visit for asthma, hospitalization or ICU stay for asthma, 3 days in succession of doubling use of SABA or need for systemic steroids if not on systemic steroids, or increase of systemic steroids if normally on systemic steroid) (patient can be rescreened 4 weeks after exacerbation has resolved)
* Stable lung function, reduction in no more than 20% (or clinically significant per patient) reduction of pulmonary function testing from time of stability
* History of being seen or had intervention/care based upon evaluation in Functional Medicine Institute or following Functional Medicine principles/ approach to asthma care.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2020-05 (Actual); Study Completion 2021-02 (Actual)

PRIMARY OUTCOMES:
Asthma Control | 9 Months
  Measured by Asthma Control Test Questionnaire (ACQ)
Asthma Control | 9 Months
  Measured by Asthma Quality of Life Questionnaire (AQLQ)

SECONDARY OUTCOMES:
Measurement of Airflow | 9 Months
  Spirometry measures of forced expiratory volume at one second (FEV1) and forced vital capacity (FVC)
Measurement of Airflow | 9 Months
  Bronchodilator response, specific airway conductance (% SGaw) and specific airway resistance (SRaw)
Daily Variability in Airflow | 9 Months
  Peak flow measured twice daily and recorded in a diary
Noninvasive Markers of Airway Inflammation | 9 months
  Measurement of exhaled Nitric Oxide
Quantity of Controller Medications Needed for Stability | 9 months
  Total inhaled corticosteroid (ICS) dose

CONTACTS AND LOCATIONS:
Overall Officials: Sumita Khatri, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- The Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No